CLINICAL TRIAL: NCT01626417
Title: A Prospective, Experimental Study to Evaluate Transfer Kinematics and Kinetics of Chronic Post-stroke Patients With Tibion Bionic Leg
Brief Title: Evaluation of Transfer Kinematics and Kinetics in Patients Chronic Post-stroke Using the Tibion Bionic Leg
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tibion Bionics, Inc. (Industry)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CP 007
Record Dates: First submitted 2012-06-18; First posted 2012-06-22 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Stroke
Keywords: Stroke; Tibion; Bionics; Rehab; Therapy; Robotics; Intention
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient Population (No Intervention): Chronic post-stroke subjects with varied impairment level, who have completed routine rehabilitative physical therapy.
  Interventions: Device: Tibion Bionic Leg

INTERVENTIONS:
Device: Tibion Bionic Leg — The device is a lightweight, wearable, portable, battery-powered, robotic leg orthosis that provides active assistance and resistance to lower limb movement according to the patient's intent to move.

SUMMARY:
The objective of this clinical study is to examine the acute kinematics and kinetics of utilizing the Tibion Bionic Leg in a sample of chronic post-stroke patients performing sit-to-stand and stand-to-sit transfers across a range of assistance and resistance settings (internal to the device); to compare these metrics to baseline performance without the Bionic Leg; and to determine the Bionic Leg settings that optimize a restorative (equal force distribution) movement state in these patients.

DETAILED DESCRIPTION:
Comprehensive motion (kinetics and kinematics) data specific to sit-to-stand and stand-to-sit transfers with and without the Tibion Bionic Leg. The Vicon Motion Analysis System will be utilized to track movement using markers on the subject and the Bionic Leg per the UCSF Human Performance Center's routine. Once outfitted with the marker system, patients will be instructed to perform multiple sit-to-stand and stand-to-sit transfers while data is gathered.

The sit-to-stand and stand-to-sit transfers will be performed using a standard chair, with a seat height not less than 12" from the floor. The chair will be positioned such that, at sitting rest, each of the subject's feet are positioned on limb-specific force plates (left and right).

ELIGIBILITY:
Inclusion Criteria:

* Single ischemic stroke with residual unilateral lower-extremity weakness
* Chronic post-stroke (>12 months since event)
* Eligible to participate to lower extremity physical therapy
* Age 30 years or greater
* Able to ambulate at least 10 meters without therapist assistance
* Able to ambulate without a leg brace
* Able to transfer from sitting to standing without physical assistance from a therapist
* Able to transfer from standing to sitting without physical assistance from a therapist
* Subject must understand the nature of the study and provide written informed consent prior to enrollment.
* Subject must be willing and able to attend all study sessions

Exclusion Criteria:

* Medically unstable
* Age younger than 30 years
* Subacute post-stroke (< 12 months since event)
* Status-post multiple strokes
* Status-post traumatic brain injury
* Not eligible to participate in lower extremity physical therapy
* Concomitant degenerative neurological conditions
* Not able to ambulate at least 10 meters without therapist assistance
* Unable to ambulate without a leg brace
* Unable to transfer from sitting to standing without physical assistance from a therapist
* Unable to transfer from standing to sitting without physical assistance from a therapist
* Unable to follow instructions, complete follow-up, or provide informed consent.
* Currently enrolled in another investigational device or drug trial

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Force | Subject participation in the study is up to one (1) week.
  Force, in Newtons (N), by limb, as measured by kinematic and kinetic analysis during sit-to-stand and stand-to-sit transfers with and without the Tibion Bionic Leg.

SECONDARY OUTCOMES:
Work | Subject participation in study is up to one (1) week.
  Work, in Joules (J), by limb, as measured by kinematic and kinetic analysis during sit-to-stand and stand-to-sit transfers with and without the Tibion Bionic Leg.
Torque | Subject participation is up to one (1) week
  Torque, in Newton-meters (N-m), at the ankle and knee, by limb, as measured by kinematic and kinetic analysis during sit-to-stand and stand-to-sit transfers with and without the Tibion Bionic Leg.
Moment | Subject participation is up to one (1) week
  Moment at the ankle and knee in Newtons (N), by limb, as measured by kinematic and kinetic analysis during sit-to-stand and stand-to-sit transfers with and without the Tibion Bionic Leg.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua G Vose, MD, Principal Investigator — Tibion Corporation
Locations (2):
- United States (2):
  - UCSF Human Performance Center, San Francisco, California
  - Tibion Corporation, Sunnyvale, California

REFERENCES:
- [Background] Wong CK, Bishop L, Stein J. A wearable robotic knee orthosis for gait training: a case-series of hemiparetic stroke survivors. Prosthet Orthot Int. 2012 Mar;36(1):113-20. doi: 10.1177/0309364611428235. Epub 2011 Nov 14. PMID 22082495
- [Background] Horst RW. A bio-robotic leg orthosis for rehabilitation and mobility enhancement. Annu Int Conf IEEE Eng Med Biol Soc. 2009;2009:5030-3. doi: 10.1109/IEMBS.2009.5333581. PMID 19964374
- [Background] Horst RW, Marcus RR. FlexCVA: a continuously variable actuator for active orthotics. Conf Proc IEEE Eng Med Biol Soc. 2006;2006:2425-8. doi: 10.1109/IEMBS.2006.259950. PMID 17946511
- See also: Tibion Bionic Leg — http://www.Tibion.com